CLINICAL TRIAL: NCT03134989
Title: Association Between Intra-Operative Cochlear Response Telemetry and Hearing Preservation
Brief Title: Cochlear Response Telemetry and Hearing Preservation
Acronym: CREST
Status: Terminated | Type: Interventional
Why Stopped: slow enrolment
Sponsor: Cochlear (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CLTD5667
Record Dates: First submitted 2017-04-19; First posted 2017-05-01 (Actual); Results first posted 2021-09-24 (Actual); Last update posted 2021-09-24 (Actual); Status verified 2021-08

CONDITIONS: Hearing Impairment, Sensorineural
Keywords: cochlear implantation, electrocochleography
MeSH Terms: conditions — Hearing Loss, Sensorineural | interventions — Cochlear Implants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | Unapproved Device: Yes

ARMS (1):
- Cochlear implant recipients (Other): Study group is comprised of cochlear implant patients already identified as candidates and undergoing surgery.
  Interventions: Device: Cochlear implant

INTERVENTIONS:
Device: Cochlear implant — Study involves measuring using Electrocochleography to measure the CM response in patients undergoing cochlear implant surgery

SUMMARY:
The main purpose of this study is to monitor the response from the cochlea as the electrode is inserted during the operation to receive a cochlear implant. The Cochlear Response Telemetry tool aims to measure the response from the cells within the cochlea and may be useful in the future to help to improve the surgical technique and potentially help surgeons better preserve any natural hearing that is available. The measurements are obtained using the cochlear implant and sound processor while a sound is presented to the ear through an earphone (like an earplug) placed into the ear canal.

ELIGIBILITY:
Inclusion Criteria:

* Candidate for cochlear implantation (with CI522, CI532, CI622, CI632 or Hybrid-L24 (US only) according to local indications
* 18 years of age or older at the time of enrolment
* Pre-operative audiometric threshold in the implanted ear at 500 Hz of better than or equal to 80 dB HL
* Willingness to participate in and to comply with all requirements of the protocol

Exclusion Criteria:

* Prior cochlear implantation in the ear to be implanted
* Ossification or any other cochlear anomaly that might prevent complete insertion of the electrode array
* Abnormal cochlear/nerve anatomy on pre-operative CT or MRI imaging (excluding a mild Mondini malformation or Large Vestibular Aqueduct Syndrome)
* Deafness due to lesions of the acoustic nerve or central auditory pathway
* Diagnosis of auditory neuropathy
* Active middle-ear infection
* Additional handicaps that would prevent participation in evaluations
* Unrealistic expectations on the part of the subject, regarding the possible benefits, risks and limitations that are inherent to the procedure and investigational device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2017-12-22 (Actual); Primary Completion 2020-06-18 (Actual); Study Completion 2020-06-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Italiano de Buenos Aires, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Adults Implanted With CI522, CI532, CI622, CI632 or Hybrid-L24 (US Only): Adults (≥ 18 years of age) implanted with CI522, CI532, CI622, CI632 or Hybrid-L24 (US only) with pre-operative audiometric threshold in the ear to be implanted of better than or equal to 80 dB HL at the frequency of 500 Hz.
Period: Overall Study
Arm/Group | Adults Implanted With CI522, CI532, CI622, CI632 or Hybrid-L24 (US Only)
Started | 80
Completed | 80 (Clinical investigation termination date: Last Subject, Final Visit 18-Jun-2020)
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 19 data points were excluded from the analysis due to a number of reasons (outlined in the CIR), including that surgical intervention occurred during ECochG measurement for 3 patients invalidating the measures, ECochG measures were not captured intraoperatively for 5 patients, 3 patients received CI512 cochlear implant, one patient unable to undergo surgery, 7 patients had issues with the audiometric measurements.
Arm/Group | Adults Implanted With CI522, CI532, CI622, CI632 or Hybrid-L24 (US Only)
Number analyzed (Participants) | 61
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 36
  >=65 years | 25
Age, Continuous [Mean (Full Range); unit: Years] | 59.7 [19 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 26
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Device [Number; unit: participants]
  CI522/522 | 52
  CI532 | 9
AETIOLOGY [Number; unit: participants]
  Unknown | 39
  Otosclerosis | 2
  Genetic | 8
  Meniere's Disease | 1
  Sudden Hearing Loss | 2
  Chronic Otitis Media | 1
  Usher's Syndrome | 3
  DeaFNess Autosomal Dominant 9 (DFNA9) | 1
  Noise Exposure | 4
EAR (Left/Right [Number; unit: participants]
  Left Ear | 31
  Right Ear | 30
Nature of Hearing loss [Number; unit: participants]
  PROGRESSIVE | 47
  CONGENITAL WITH PROGRESSION | 8
  SUDDEN | 4
  PROGRESSION WITH SUDDEN | 1
  No Data | 1
Age of onset of hearing loss [Mean (Full Range); unit: Years] — Population: No data from one patient in this study
  Years
    number analyzed (Participants) | 60
    (all) | 30.75 [0 to 70]
Age of diagnosis Severe -Profound Hearing Loss [Mean (Full Range); unit: Years] — Population: Total Analysis population=61 Subjects with No diagnosis=9 Subjects with No data =1
  Hence, Measure Analysis Population=51
  Years
    number analyzed (Participants) | 51
    (all) | 46.98 [0 to 83]

OUTCOME MEASURES:

1. Primary Outcome: Change in Low-frequency Hearing Thresholds Assessed Audiometrically Pre- and Post-operatively.
Description: Average low-frequency (LF) hearing thresholds (average thresholds at 500, 750, and 1000 Hz) will be measured for the implanted ear 4 to 6 weeks following surgery and compared with average LF hearing thresholds measured relative to the pre-operative baseline measured within 90 days of CI surgery. The outcome measure of interest is the change in average LF hearing thresholds pre- to postoperative for each subject. The average change observed for individual subjects will then be compared with individual electrophysiological cochlear microphonic (CM) measures made during the surgery using the Cochlear Response Telemetry System. Of specific interest is whether or not compromised CM measures relate to pre-to-postoperative changes in low-frequency hearing. In other words, are larger changes in average LF hearing thresholds observed in subjects with compromised CM measures made intraoperative versus those with uncompromised CM response?
Time Frame: Baseline measurement (pre-operatively) compared to 4 to 6 weeks post-surgery
Population: 19 of the 80 ECochG intro-operative responses were excluded from the analysis (reasons are outlined in the CIR). A further 18 of the remaining 61 data points were excluded due to an unclear CM response resulting in N=43 responses categorized as either preserved or compromised. Further, two subjects were excluded from the primary endpoint analysis as there were no FUV1 thresholds collected. Thereby N=41.
Measure: Mean (Full Range); unit: dB
Groups:
- Cochlear Implant Recipients: Study group is comprised of cochlear implant patients already identified as candidates and undergoing surgery.
  Cochlear implant: Study involves using Electrocochleography to measure the CM response in patients undergoing cochlear implant surgery
Arm/Group | Cochlear Implant Recipients
Number analyzed (Participants) | 41
dB | 26.9 [15 to 60]

2. Secondary Outcome: Change in Low-frequency Hearing Thresholds Assessed Audiometrically Pre- and Post-operatively.
Description: Average low-frequency (LF) hearing thresholds (average thresholds at 500, 750, and 1000 Hz) will be measured for the implanted ear 3 months following cochlear implant activation and compared with average LF hearing thresholds measured preoperatively. The outcome measure of interest is the change in average LF hearing thresholds pre- to postoperative for each subject. The average change observed for individual subjects will then be compared with individual electrophysiological cochlear microphonic (CM) measures made during the surgery using the Cochlear Response Telemetry System. Of specific interest is whether or not compromised CM measures relate to pre-to-postoperative changes in low-frequency hearing. In other words, are larger changes in average LF hearing thresholds observed in subjects with compromised CM measures made intraoperative versus those with uncompromised CM response.
Time Frame: Baseline (pre-operative) compared to 3 months post cochlear implant activation
Population: 5 data points were excluded from this analysis due to post-operative thresholds not being measured at FUV2 (43 - 5 = 38).
Measure: Mean (Full Range); unit: dB
Arm/Group | Cochlear Implant Recipients
Number analyzed (Participants) | 38
dB | 31.52 [0 to 60]

3. Secondary Outcome: Correlation of Preoperative High-frequency Hearing Thresholds and Cochlear Microphonic Response (Number of Electrodes Inserted When CM Detected).
Description: The onset of the cochlear microphonic (CM) response will be measured intraoperative to determine if there is a relationship between the onset of the CM response during electrode insertion and the preoperative high-frequency acoustic hearing thresholds. The onset of the CM response will be tracked by impedance measures that are interleaved with the CM recordings. As each electrode in the array enters the perilymph in the cochlea there will be a measured reduction in impedance. CM onset will be defined in terms of the nth electrode (out of the 22 electrodes) to enter the cochlea. Preoperative high-frequency hearing will be defined as the average of preoperative thresholds at frequencies of 2 kHz, 3 kHz and 4 kHz for each individual subject.
Time Frame: Intraoperative
Population: 40 data points with a CM response were eligible to be analysed for this outcome. Those excluded were due to an absence of CM under visual inspection (n =16), an absence of the impedance measurement used to calculate depth (n = 4), or an array that was withdrawn or reinserted at any time (n = 5).
Measure: Number; unit: Pearson correlation coefficient
Groups:
- Cochlear Implant Recipients: Study group is comprised of cochlear implant patients already identified as candidates and undergoing surgery.
  Cochlear implant: Study involves Electrocochleography to measure the CM response in patients undergoing cochlear implant surgery
Arm/Group | Cochlear Implant Recipients
Number analyzed (Participants) | 40
Pearson correlation coefficient | 0.78

ADVERSE EVENTS:
Time Frame: 5 months
Description: Adverse events were collected for the subjects duration of involvement in the study - which was expected to be 5 months
Groups:
- Cochlear Implant Recipients: Study group is comprised of cochlear implant patients already identified as candidates and undergoing surgery.
  Cochlear implant: Study involves measuring cochlear response electrophysiologically during surgery to place a cochlear implant in patients already identified as candidates.
Arm/Group | Cochlear Implant Recipients
All-Cause Mortality (participants affected / at risk) | 0/61
Serious Adverse Events (participants affected / at risk) | 2/61
Other Adverse Events (participants affected / at risk) | 15/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cochlear Implant Recipients (N=61)
SUDDEN ONSET ROTARY VERTIGO (Surgical and medical procedures) | 2 — PATIENT EXPERIENCED DIZZINESS, NAUSEA AND VOMITING AFTER POST-OP STENVERS X-RAY PROCEDURE DUE TO MANIPULATION TO GET GOOD IMAGE. DIZZINESS SETTLED AFTER ABOUT 1 HOUR. NAUSEA MAY BE RELATED TO CLINDAMYCIN POST-OP DOSE, DOSAGE CORRECTED.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cochlear Implant Recipients (N=61)
COLD (General disorders) | 1 (1)
UNDISPLACED FRACTURE OF THE MEDIAL FEMORAL CONDYLE (Musculoskeletal and connective tissue disorders) | 1 (1)
DELAYED FACIAL PARALYSIS (Musculoskeletal and connective tissue disorders) | 1 (1)
VERTIGO AND NAUSEA (General disorders) | 4 (4)
BRONCHITIS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTITIS MEDIA WITH EFFUSION (Ear and labyrinth disorders) | 1 (1)
OTITIS EXTERNA DURING SURGERY (Ear and labyrinth disorders) | 1 (1)
INTRAOPERATIVE HORIZONTAL CANAL DEFECT resulted in 'SEVERE VERTIGO EXPERIENCED DURING AUDIOMETRY, TY (General disorders) | 1 (1)
PULSATILE TINNITUS (Ear and labyrinth disorders) | 1 (1)
PAIN AND INFLAMATION POST SURGERY (Ear and labyrinth disorders) | 1 (1)
EXACERBATION MENIERE'S DISEASE (Ear and labyrinth disorders) | 1 (1)
BLOOD/FLUID STILL BEHIND EAR; NO PAIN REPORTED BY PATIENT (Ear and labyrinth disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-08-23): https://cdn.clinicaltrials.gov/large-docs/89/NCT03134989/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-29): https://cdn.clinicaltrials.gov/large-docs/89/NCT03134989/SAP_001.pdf